CLINICAL TRIAL: NCT01800344
Title: The Effect of a New Supraglottic Airway With Built-in Cuff Pressure Indicator on Postoperative Pharyngolaryngeal Adverse Events: A Prospective, Randomized Trial
Brief Title: The Effect of a New Supraglottic Airway With Built-in Cuff Pressure Indicator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 11-0392-A
Record Dates: First submitted 2013-02-08; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: The Study Focuses on the Effect of a New Supraglottic Airway With Built-in Cuff Pressure Indicator on Postoperative Pharyngolaryngeal Adverse Events
Keywords: Airway Cuff; LMA; Ultra; Cuff Pressure; Ventilation; Anesthesia; Intubation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The laryngeal mask airway-ClassicTM (LMA) (Active Comparator): The LMA is a large foreign body that exerts pressure on the pharyngeal mucosa. High LMA intracuff pressures may reduce pharyngeal mucosal perfusion and lead to throat discomfort.
  Interventions: Device: LMA
- The AES Ultra CPVTM LMA (Ultra) (Active Comparator): Ultra is a new supraglottic airway with anatomical features and insertion technique virtually identical to the LMA-ClassicTM. The cuff and the shaft are made of silicone with a built-in CPV pilot balloon valve which provides continuous monitoring of the intracuff pressure. The CPV cuff pressure indicator has 3 zones indicated by color: yellow corresponds to pressure < 50 cm H2O; green 60 cm H2O; and red >70 cm H2O
  Interventions: Device: Ultra

INTERVENTIONS:
Device: LMA
  Other Names: The laryngeal mask airway-Classic
  Arms: The laryngeal mask airway-ClassicTM (LMA)
Device: Ultra — Ultra
  Other Names: AES Ultra CPVTM LMA (Ultra)
  Arms: The AES Ultra CPVTM LMA (Ultra)

SUMMARY:
The study compares the incidence of pharyngolaryngeal complications in patients managed with either a pressure-limiting strategy using the AES Ultra CPVTM or a standard practice using a LMA, in ambulatory surgery patients.

DETAILED DESCRIPTION:
Recent evidence suggests that reduction of LMA intracuff pressure may decrease the incidence of pharyngolaryngeal symptoms. Yet, pressure manometers are not widely available limiting the application of a strategy of intracuff pressure reduction. The Ultra airway has been designed to provide continuous indication of intracuff pressure and can limit the intracuff pressure to < 60 cm H2O. This study compares the incidence of pharyngolaryngeal complications in patients managed with either a pressure-limiting strategy using the Ultra or a standard practice using a LMA, in ambulatory surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I-III
* 18 to 65 years of age
* Ambulatory patients scheduled to undergo knee arthroscopy, transurethral resection of bladder tumor, hand, gynecological, general surgical and eye procedures under a short general anesthesia of less than 2 hours
* Spontaneously breathing on the LMA

Exclusion Criteria:

* Reduced mouth opening less than 2.5cm
* Recent history of upper respiratory tract infection and sore throats
* Contraindications of LMA use (Morbid obesity with body mass index greater than 40kg/m2, symptomatic hiatus hernia, esophageal reflux disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome, composite pharyngolaryngeal complication, is defined as the presence of either sore throat, dysphonia or dysphagia at 1, 2, and 24 h postoperatively. | 1, 2, 24 hours

SECONDARY OUTCOMES:
Intracuff pressure | intraoperative
  Intracuff pressure intraoperative 10 post insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Health Network- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wong DT, Tam AD, Mehta V, Raveendran R, Riad W, Chung FF. New supraglottic airway with built-in pressure indicator decreases postoperative pharyngolaryngeal symptoms: a randomized controlled trial. Can J Anaesth. 2013 Dec;60(12):1197-203. doi: 10.1007/s12630-013-0044-2. Epub 2013 Oct 5. PMID 24097301